CLINICAL TRIAL: NCT01677702
Title: The Clinical Research on the Efficiency of Yili Lactoferrin Shuhua Milk in the Improvement of Human Immunization
Brief Title: Study of Yili Lactoferrin ShuHua Milk in the Improvement of Human Immunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Yili Industrial Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YL/CL-002
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Immunization; Human Influenza; Common Cold
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — Lactoferrin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Yili Lactoferrin ShuHua Milk (lactoferrin 5mg/100ml) (Active Comparator): Total 250mL milk (with lactoferrin 5mg/100ml) will be taken once per day at 10am daily during the 84 days intervention.
  Interventions: Dietary Supplement: Yili Lactoferrin ShuHua Milk (Lactoferrin 5mg/100ml)
- Yili Lactoferrin ShuHua Milk (lactoferrin 10mg/100ml) (Active Comparator): Total 250mL milk (with lactoferrin 10mg/100ml) will be taken once per day at 10am daily during the 84 days intervention.
  Interventions: Dietary Supplement: Yili Lactoferrin ShuHua Milk (Lactoferrin 10mg/100ml)
- Recombined low-protein milk (Placebo Comparator): Total 250mL placebo milk will be taken once per day at 10am daily during the 84 days intervention.
  Interventions: Dietary Supplement: Recombined low protein milk

INTERVENTIONS:
Dietary Supplement: Yili Lactoferrin ShuHua Milk (Lactoferrin 5mg/100ml) — Total 250mL milk (with lactoferrin 5mg/100ml) will be taken once per day at 10am daily during the 84 days intervention.
  Arms: Yili Lactoferrin ShuHua Milk (lactoferrin 5mg/100ml)
Dietary Supplement: Yili Lactoferrin ShuHua Milk (Lactoferrin 10mg/100ml) — Total 250mL milk (with lactoferrin 10mg/100ml) will be taken once per day at 10am daily during the 84 days intervention.
  Arms: Yili Lactoferrin ShuHua Milk (lactoferrin 10mg/100ml)
Dietary Supplement: Recombined low protein milk — Total 250ml of placebo milk will be taken once a day at 10am daily during the 84 day intervention.
  Arms: Recombined low-protein milk

SUMMARY:
The purpose of this study is to determine whether Yili Lactoferrin ShuHua Milk are effective in reducing the occurrence of flu symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years, catch cold for 4 to 6 times in last year;
* Age 35 to 45 years, catch cold for 4 to 6 times in recent 3 month;
* Age 60 to 75 years, catch cold for 4 to 6 times in last year;
* BMI 18.5to 29.9kg/m2;
* Able to understand the nature and purpose of the study including potential risks and side effects

Exclusion Criteria:

* Recent (within 6 months of screening) been vaccinated influenza vaccine, or recent (within 15 days of screening) been vaccinated ther vaccines;
* Suffering from rhinitis chronic, laryngitis, labored breathing that similar to flu symptoms. Such as chronic allergic rhinitis, asthma, COPD;
* Long-term use of any prescription or OTC medication that inhibit or prevent flu symptoms, including but not limited to, antihistamine, pectoral, high doses of vitamin C;
* Recent use (within 3 months of screening) of any prescription or OTC medication that significantly affects immune response, such as antibiotic;
* Known allergies to dairy and any substance in the study product;
* History of alcohol, drug, or medication abuse
* Pregnant or breastfeeding women
* Recent daily use (within 3 months of screening) of any probiotics, clabber or yogurt;
* Any comorbidity that could, in the opinion of the investigator, preclude the subject's ability to successfully and safely complete the study or that may confound study outcomes

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Assess occurrence of flu symptoms during intervention | 3 months

SECONDARY OUTCOMES:
Assess severity of flu symptoms | 3 months
Proportion of subjects which require treatment with flu medication | 3 months
Change in immune markers such as antibodies and interleukins | Baseline & 3 months
Record subject sick leave due to flu | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ying An, Ph.D, Study Director — Inner Mongolia Hilo Industrial Group Co., Ltd; Donglian Cai, Principal Investigator — Changhai Hospital of Shanghai, Nutriology Dept.; Yeqing Shi, Principal Investigator — Changhai Hospital of Shanghai, Rheumatology Dept.
Locations (2):
- China (2):
  - NanMoFang Community Health Service Center, Chao Yang District, Beijing Municipality
  - JuQuan Community Health Service Center, GuCun, Baoshan District,, Shanghai Municipality